CLINICAL TRIAL: NCT04636476
Title: One Stage Correction of Congenital Penile Curvature Complex
Acronym: Al-AzharCPCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: dr. Muhammad Abdelhafez Mahmoud, MD (Other)
Responsible Party: Sponsor-Investigator, dr. Muhammad Abdelhafez Mahmoud, MD, Lecturer of pediatric surgery, Al-Azhar university, Faculty of Medicine, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Al-AzharCPCC
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Congenital Anomaly; Chordee; Curvature of Penis; Torsion of the Penis
Keywords: Congenital penile curvature;; Penile rotation;; Dorsal dartos flap;; Complex anomaly
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Intervention Model Description: Sequential Assignment Prospective cohort study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Modified Nesbit technique followed by dorsal dartos flap (Other): Modified Nesbit technique to correct penile curvature followed by dorsal dartos flap to correct penile torsion
  Interventions: Procedure: Modified Nesbit's procedure and dorsal dartos flap

INTERVENTIONS:
Procedure: Modified Nesbit's procedure and dorsal dartos flap — Modified Nesbit's procedure to correct the penile curvature and dorsal dartos flap to correct the associated penile torsion

SUMMARY:
To present update & experience in management of congenital penile curvature complex.

DETAILED DESCRIPTION:
Type of study: prospective study

Review of literature:

* Different modalities of urethroplasty for correction of CPCC without hypospadias (Nesbit, modified Nesbit, dorsal dartos flap, combined plication-incision CPI, suture fixation to pubic bone).
* Merits of modified Nesbit technique accompanied by dorsal dartos flap for one-stage correction of CPCC without hypospadias.

This is a prospective study conducted at pediatric surgery department, New Damietta & Alhoussain Al-Azhar University Hospitals, from January 2015 to May 2020, on 56 male patients with isolated CPCC. All of them will undergo one-stage correction corporoplasty using modified Nesbit technique accompanied by dorsal dartos flap.

Institutes of the study:

A multicenter study at Pediatric Surgery Departments, Al-Azhar University hospitals at New Damietta & Cairo. Number of cases: Fifty-six male patients. Time frame: period of 5.6 years.

Ethical Consideration:

The protocol will be discussed and approved for clinical study by the Ethical Research Committee at the principal investigator's hospital. The study protocol was approved by local research and ethics committee of Al-Azhar Faculty of Medicine; the study protocol was explained to all guardians and their informed consents were obtained for involvement in the study. Confidentiality and the right to withdraw from the study at any time were guaranteed.

Preoperative preparation:

Children with CPCC those fulfill inclusion criteria will undergo a nursing evaluation of functional health status and a preoperative evaluation by an anesthesiologist & pediatrician. The angle of penile rotation will be measured on the photograph, using Millen Med DICOM viewer program for image analysis, based on the orientation of the urethral meatus relative to the vertical position.

Follow-up:

Patients will be followed-up at OPD.

Statistical Analysis:

Data will be summarized into continuous variables expressed as mean ± standard deviation and categorical variables expressed as frequency count and percentage (%), using appropriate software computer package. Fisher's exact test is used for comparison of frequency counts/percentage. A two-sided p-value < 0.05 is considered statistically significant.

Discussion:

It will focus on one-stage correction of congenital penile curvature complex (CPCC) using modified Nesbit's procedure (to correct curvature) and dorsal dartos flap (to correct torsion). The results obtained from this study will be compared between both group and with those reported in the literature. Also, it will focus on results, complications, their management, and clinical evaluation by noticing urine stream direction. At the end, the investigators will conclude that this technique ensures correction of the complex penile anomaly with satisfactory results and nice cosmetic outcome.

ELIGIBILITY:
Inclusion Criteria:

* 2 to 10 years old boys
* with congenital curvature complex of the penis
* with normally situated urethral meatus.
* The various degrees of penile curvature ranged between 30° - 90° associated with 30° - 90° penile rotation

Exclusion Criteria:

* Boys with CPCC with abnormal urethral meatus as hypospadias or epispadias, or
* with the range of angle degree of penile curvature less than 30° associated with less than 30° penile rotation or
* with acquired penile curvature or
* having an isolated lesion.

Ages: 2 Years to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Male children from 2-10 years old with CPCC with normal urethral meatus
Enrollment: 56 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Clockwise rotation | 5 years
  Clockwise rotation of the penis (number & percent)
Counterlockwise rotation | 5 years
  Counterlockwise rotation of the penis (number & percent)
Ventral Curvature | 5 years
  Ventral Curvature of the penis (number & percent)
Dorsal Curvature | 5 years
  Dorsal Curvature of the penis (number & percent)
Lateral Curvature | 5 years
  Lateral Curvature of the penis (number & percent)
Age | 5 years
  Age of the patients (years)
Operative time | 1 day (day of surgery)
  Operative time (minutes)
Post-operative hospital stay | 1 week
  Hospital stay period (days)
Post-operative follow-up period | 5 years
  Follow-up period (months)

SECONDARY OUTCOMES:
Functional impairment | 5 years
  Functional impairment (number & percent)
Aesthetic impairment | 5 years
  Aesthetic impairment (number & percent)
Residual curvature > 10° | 5 years
  Residual curvature > 10° (number & percent)
Residual rotation > 10° | 5 years
  Residual rotation > 10° (number & percent)
Post-operative paresthesia | 5 years
  Post-operative paresthesia (number & percent)
Skin ischemia | 5 years
  Skin ischemia (number & percent)
Hematoma | 5 years
  Hematoma (number & percent)
Dressing soaked with blood | 5 years
  Dressing soaked with blood (number & percent)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M Shahin, MD,PhD, Principal Investigator — Al-Azhar New Damietta University
Locations (1):
- Mohamed M Shahin, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data will be available for other researchers including methodology, figures, tables, results, and philosophy of discussion and the value this study will add to the literature
Supporting Information: Study Protocol, SAP, ICF
Time Frame: from now indefinitely
Access Criteria: after the article became accepted and available online.